CLINICAL TRIAL: NCT01967589
Title: Investigation on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of a Long Acting GLP-1 Analogue (NNC0113-0987) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9926-3950; 2012-002893-30 (EudraCT Number); U1111-1131-8724 (Other: WHO)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- DC (dosing condition) (Experimental): Escalation design.
  Interventions: Drug: NNC0113-0987; Drug: placebo
- Oral A (Experimental): Escalation design. Planned end-dose is 5 mg.
  Interventions: Drug: NNC0113-0987; Drug: placebo
- Oral B (Experimental): Escalation design. Planned end-dose is 10 mg.
  Interventions: Drug: NNC0113-0987; Drug: placebo
- Oral C (Experimental): Escalation design. Planned end-dose is 20 mg.
  Interventions: Drug: NNC0113-0987; Drug: placebo

INTERVENTIONS:
Drug: NNC0113-0987 — Once-daily doses for oral administration. Multiple doses with sequential dose increments over 10 weeks. Progression to next dose increment is based on a safety evaluation
Drug: placebo — Once-daily doses for oral administration

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of multiple doses of a long acting GLP-1 analogue (NNC0113-0987) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male, who is considered to be generally healthy, based on the medical history, physical examination and the results of vital signs, electrocardiogram (ECG) and laboratory safety tests performed during the screening visit, as judged by the investigator
* Age 18-64 years (both inclusive) at the time of signing informed consent
* BMI (body mass index) 20.0-29.9 kg/m^2 (both inclusive)

Exclusion Criteria:

* History of, or presence of, cancer, diabetes or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal (GI), endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders, as judged by the investigator
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Use of prescription or non-prescription medicinal and herbal products (except routine vitamins) within three weeks preceding the dosing period. Occasional use of paracetamol or acetylsalicylic acid is permitted
* Subject with previous GI surgery, except subjects that underwent uncomplicated surgical procedures such as appendectomy, hernia surgery, biopsies, as well as colonic and gastric endoscopy

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) recorded | From the time of first dosing (Day 0) and until completion of the post-treatment follow-up visit (Day 83-97)

SECONDARY OUTCOMES:
Area under the NNC0113-0987 plasma concentration curve | During a dosing interval (0-24 hours) at steady state (Day 67; Day 68 and Day 69)
Maximum observed NNC0113-0987 plasma concentration | During a dosing interval (0-24 hours) at steady state (Day 67; Day 68 and Day 69)
Time to maximum observed NNC0113-0987 plasma concentration | During a dosing interval (0-24 hours) at steady state (Day 67; Day 68 and Day 69)
Change in fasting plasma glucose (FPG) | From baseline (Day 0, pre-dose) to after 10 weeks of treatment (Day 70)
Change in HbA1C (glycosylated haemoglobin) | From baseline (Day 0, pre-dose) to after 10 weeks of treatment (Day 70)
Change in body weight | From baseline (Day -1) to after 10 weeks of treatment (Day 70)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Harrow, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com